CLINICAL TRIAL: NCT00461669
Title: Hip Fracture Characterization With Ultrasound Exam
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Other Study IDs: HIPUS-2
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-03

CONDITIONS: Hip Fractures
Keywords: hip; fracture; ultrasound
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ultrasound examination of the hip

SUMMARY:
Hip fractures are usually classified according to their X-ray as subcapital, pertrochanteric. We examine hip fractures with ultrasound in order to characterize the fractures with several parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients over 50 years with x rays showing a hip fracture

Exclusion Criteria:

* previous fracture or surgical intervention in the hip
* fracture over 3 days old
* pregnancy
* flexion contracture of hip

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Alon Burg, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel